CLINICAL TRIAL: NCT04737941
Title: Finnish Venous Ulcer Study
Brief Title: Finnish Venous Ulcer Study (FINNULCER Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Toni Pihlaja, Principal Investigator, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/2021
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Venous Leg Ulcer
Keywords: Venous Leg Ulcer; Foam Sclerotherapy; Endothermal Ablation; Sub-ulcer Foam Sclerotherapy
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First-visit foam sclerotherapy (Experimental): Patients in the first-visit foam sclerotherapy group undergo first-visit foam sclerotherapy (including sub-ulcer foam sclerotherapy), and truncal vein endothermal ablation is scheduled when the anatomy is suitable. Compression therapy is initiated immediately.
  Interventions: Procedure: Endothermal Ablation; Procedure: Foam Sclerotherapy
- Scheduled treatment (Active Comparator): Patients in the scheduled treatment group receive scheduled endovenous ablation, including foam sclerotherapy and/or endothermal ablation, depending on reflux anatomy. This group represents the current standard of care. Compression therapy is initiated immediately.
  Interventions: Procedure: Endothermal Ablation; Procedure: Foam Sclerotherapy

INTERVENTIONS:
Procedure: Endothermal Ablation — Endothermal ablation is performed to suitable insufficient truncal veins (Great-, Anterior Accessory- and/or Small Saphenous Vein)
Procedure: Foam Sclerotherapy — Foam sclerotherapy is performed to insufficient veins distal to the truncal superficial veins.

SUMMARY:
This multicenter randomized controlled trial evaluates the effect of first-visit foam sclerotherapy (including sub-ulcer foam sclerotherapy) in patients with venous leg ulcer.

DETAILED DESCRIPTION:
To evaluate the effect of first-visit foam sclerotherapy, patients with venous leg ulcers are randomly assigned to either the first-visit foam sclerotherapy group or the scheduled treatment group. The scheduled treatment group represents the current standard of care. The primary outcome of this study is the time to ulcer healing.

In addition to the first-visit treatment in the study group, both groups receive endothermal ablation and/or foam sclerotherapy to (further) treat ulcer-related insufficient veins and truncal insufficiency in scheduled treatment visit(s).

Class 2 thigh-high compression or the best possible compression therapy tolerated by the patient is provided in both groups. The follow-up period for the primary outcome is one year.

For this study, based on Oulu University Hospital's retrospective data (partly published in Pihlaja et al 2020) of venous ulcer healing the investigators assumed Hazard Ratio 1.5 for venous ulcer to heal in first-visit foam sclerotherapy group compared to scheduled treatment group.

Assuming drop-out of 10% this study recruits total of 248 patients (a=0.05, b=0.2).

ELIGIBILITY:
Inclusion Criteria:

* Patient informed consent
* Venous ulcer, aged from one month to one year
* Duplex ultrasonography verified (vein reflux greater than >0.5 second) superficial venous insufficiency
* Sufficient arterial circulation (at least on criterion met: Palpable distal pulses / ankle-brachial index > 0,8 / Toe pressure >60mmhg)

Exclusion Criteria:

* Leg ulcers other than venous etiology
* Ulcers requiring operation theater revision
* Patent foramen ovale
* Several times recurrent (over 3 recurrences) venous ulcer
* Body Mass Index over 40
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to ulcer Healing | 0-365 days
  Complete re-epithelialisation of ulcer area

SECONDARY OUTCOMES:
EQ-5D Questionnaire | 0-365 days
  Score 0-100 where higher is better
Wound-QOL Questionnaire | 0-365 days
  Score 0-17 where lower is better
Venous ulcer area | 0-365 days
  Reduction on venous ulcer maximum diameter

CONTACTS AND LOCATIONS:
Overall Officials: Toni Pihlaja, MD, Principal Investigator — Oulu University Hospital; Karoliina Halmesmaki, Docent, Principal Investigator — Helsinki University Central Hospital; Maarit Venermo, Professor, Study Chair — Helsinki University Central Hospital; Matti Pokela, Docent, Study Chair — Oulu University Hospital
Locations (5):
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Keski-Suomen keskussairaala, Jyväskylä
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa

REFERENCES:
- [Background] Pihlaja T, Torro P, Ohtonen P, Romsi P, Pokela M. Ten years of experience with first-visit foam sclerotherapy to initiate venous ulcer healing. J Vasc Surg Venous Lymphat Disord. 2021 Jul;9(4):954-960. doi: 10.1016/j.jvsv.2020.11.012. Epub 2020 Nov 25. PMID 33248300
- [Derived] Pihlaja T, Ohtonen P, Hakovirta H, Viljamaa J, Kukkonen T, Venermo M, Halmesmaki K, Pokela M. Trial protocol for evaluating sub-ulcer foam sclerotherapy as an adjunct to conventional endovenous treatment in patients with venous leg ulcers: The FINNULCER multicenter randomized controlled trial. Phlebology. 2025 Oct;40(9):713-718. doi: 10.1177/02683555251335618. Epub 2025 Apr 17. PMID 40243046